CLINICAL TRIAL: NCT04185532
Title: Treatment of Acute ACL Injuries in Young Patients Using a Rebound ACL Brace
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to problems with the brace in the majority of the patients in the treatment group; such as skin lesions, non-fitting brace and severe itching. Furthermore, half of the patients went on to ACLR.
Sponsor: Frida Hansson, MD (Other)
Responsible Party: Sponsor-Investigator, Frida Hansson, MD, MD. Principal Investigator. PhD student, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1450-31
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: ACL; children and adolescents; rebound ACL brace
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The knee laxity measurement with KT-1000 will be performed by an assessor without knowledge of type of intervention. Other outcome measures will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rebound ACL brace and physiotherapy (Experimental): The intervention will be the use of rebound ACL brace for 9 weeks, which initially is locked followed by a gradually increased range of motion. A standardized rehab protocol is applied.
  Interventions: Other: Rebound ACL brace and physioterapy
- Physiotherapy (Active Comparator): A standardized rehab protocol comparable to the experimental group but with no brace
  Interventions: Other: Physioterapy

INTERVENTIONS:
Other: Rebound ACL brace and physioterapy — Usage of rebound ACL brace and physioterapy supervised by physioterapist
  Arms: Rebound ACL brace and physiotherapy
Other: Physioterapy — Physioterapy supervised by physioterapist
  Arms: Physiotherapy

SUMMARY:
This study evaluates the use of a brace in acute anterior cruciate ligament (ACL) injuries in children and adolescents. Half of the participants will receive a so called rebound ACL brace together with a standardized rehab program supervised by a physiotherapist, while the other half will receive only the standardized rehab program supervised by a physiotherapist

DETAILED DESCRIPTION:
A well known treatment of posterior cruciate ligament injuries in the acute phase is a brace which pushes the tibia anteriorly, and the result of the treatment is often successful with healing of the ligament. Similarly, in anterior cruciate ligament injuries, it is suggested that a rebound ACL brace which pushes the tibia posteriorly can facilitate healing of the ACL. It does not have as successful treatment results as the PCL brace, but the type and location of the ACL injury has in previous studies not been well defined. We will, after having described the localisation and type of ACL injury treat the intervention group with the rebound ACL brace and a standardized rehab program and the control group with standardized rehab program alone.

The randomization is made blockwise of 4, to treatment A= Brace+physiotherapy or B=Physioterapy. The groups are stratified for gender and age (<=14 years and >14 years)

ELIGIBILITY:
Inclusion Criteria:

* No previous significant knee injury
* Trauma followed by hemarthrosis and clinical suspicion of an acute ACL injury
* Acute ACL rupture seen on MRI

Exclusion Criteria:

* Previous ipsilateral knee surgery
* Associated injuries which require early surgical intervention

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — based on self-representation of gender identity
Enrollment: 44 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Objective knee function | 6 months
  laxity measurement (KT-1000)
Objective knee function | 12 months
  laxity measurement (KT-1000)
Objective knee function | 24 months
  laxity measurement (KT-1000)
objective knee function | 6 months
  muscle strength (measured by Biodex)
objective knee function | 12 months
  muscle strength (measured by Biodex)
objective knee function | 24 months
  muscle strength (measured by Biodex)
objective knee function | 6 months
  jump tests
objective knee function | 12 months
  jump tests
objective knee function | 24 months
  jump tests

SECONDARY OUTCOMES:
Subjective knee function | 6, 12 and 24 months
  EQ-5D-Y
Subjective knee function | 6, 12 and 24 months
  The Knee injury and Osteoarthritis Outcome Score for children, KOOS child. 5 subscales, where each subscale's points are calculated to a scale from 0-100; zero representing extreme knee problems and 100 representing no knee problems
Activity level | 6, 12 and 24 months
  Presented as Tegner activity scale. The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.

CONTACTS AND LOCATIONS:
Overall Officials: Frida Hansson, MD, PhD stud, Principal Investigator — Karolinska Institutet
Locations (1):
- Capio Artro Clinic, Stockholm, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending minimum 5 years following article publication
Access Criteria: Proposals should be directed to frida.hansson@capio.se. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website
URL: https://staff.ki.se/ki-eln-the-electronic-notebook

REFERENCES:
- [Background] Jacobi M, Reischl N, Ronn K, Magnusson RA, Gautier E, Jakob RP. Healing of the Acutely Injured Anterior Cruciate Ligament: Functional Treatment with the ACL-Jack, a Dynamic Posterior Drawer Brace. Adv Orthop. 2016;2016:1609067. doi: 10.1155/2016/1609067. Epub 2016 Dec 7. PMID 28053787